CLINICAL TRIAL: NCT03985436
Title: A Pilot and Feasibility Study of a Single Session Pain Psychology Class for the Spine Surgery Patient: TREK (Transform, Restore, Empower, Knowledge) for Surgical Success
Brief Title: A Single Session Pain Psychology Class for Spine Surgery Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sara Davin, PsyD, MPH (Other)
Responsible Party: Sponsor-Investigator, Sara Davin, PsyD, MPH, Principal Investigator, The Cleveland Clinic
Organization: The Cleveland Clinic (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 19-124
Record Dates: First submitted 2019-05-03; First posted 2019-06-13 (Actual); Last update posted 2020-11-17 (Actual); Status verified 2020-11

CONDITIONS: Lumbar; Injury
MeSH Terms: conditions — Wounds and Injuries | interventions — potassium channel protein TREK-1

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Trek for Surgical Success (Experimental): Cognitive behavioral therapy for pain
  Interventions: Behavioral: Trek for Surgical Success

INTERVENTIONS:
Behavioral: Trek for Surgical Success — Cognitive behavioral therapy for pain

SUMMARY:
This project tests the feasibility a single session pain psychology class (TREK for Surgical Success) for patients undergoing spine surgery and compares outcomes in those who engage in the class to a historical group of similar patients undergoing usual care perioperatively. As of January 2020, the class option has been updated to include an online video module platform, to be used for patients unable to attend in person.

DETAILED DESCRIPTION:
The proposed study intends to utilize a psychobehavioral protocol from Darnall and colleagues to deliver a single session behavioral medicine for pain intervention for the spine surgery patient entitled "TREK (Transform, Restore, Empower, Knowledge) for Surgical Success" (TREK for SS). The intervention is based off of the above noted evidence based 2 hour pain psychology class that has been used in the chronic pain population and is also currently being tested in other surgical populations. Use of this established and evidenced based treatment for the proposed project enhances the treatment fidelity. The proposed project addresses questions in the literature such as the benefits of this class in an in-person or online format and its adaptability and effectiveness in the spine surgery population.

The primary objective of the proposed project is to determine the feasibility of a single session digital behavioral medicine for pain intervention (TREK for SS) offered the perioperative period of lumbar spine surgery as measured by patient satisfaction and intervention acceptability ratings and retention rates. In this study the perioperative period is defined as a 8 week window straddling the surgery date. A secondary objective of the study is to gather preliminary data to support the efficacy of TREK for SS as measured by relevant post surgical outcomes compared to a group of historical controls who received usual care. Should this pilot study demonstrate effectiveness in lumbar spine surgery patients, there is the potential to study larger groups of patients and to integrate the class into the standard of care as a cost-effective intervention for the spine surgery population. Additionally, findings from this pilot study could substantiate the need for training in the class protocol across disciplines so that barriers to receiving pain psychology intervention can be minimized.

ELIGIBILITY:
Inclusion Criteria:

* Adults 18 and older
* Undergoing lumbar laminectomy with or without fusion

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2019-06-10 (Actual); Primary Completion 2020-11-01 (Actual); Study Completion 2020-11-01 (Actual)

PRIMARY OUTCOMES:
Patient Satisfaction and Acceptability (change/durability of intervention acceptability) | immediately after the intervention and 12 weeks post surgery
  4 item satisfaction survey; Likert scale (1=higher acceptability of intervention for each of the 5 items; 5=least satisfaction/acceptability of the intervention) assessing acceptability of intervention; lower total score reflects higher satisfaction and acceptability
Engagement Rates of CBT-P intervention | within 2 weeks before or 2 weeks after surgery
  Class attendance
Change in Modified Oswestry Disability Index (MDQ) pre to post treatment | before surgery and 12 weeks post surgery
  Back pain-related disability, The ODI is made up of 10 questions. Each question is scored from 0-5 (minimum to maximum).The point total from each section is summed and the then divided by the total number of questions answered and multiplied by 100 to create a percentage disability. The scores range from 0-100% with lower scores meaning less disability.
Change in Pain Castastrophizing pre and post treatment | before surgery and 12 weeks post surgery
  13 item scale measuring pain catastrophizing; 5-point scales with the end points (0) not at all and (4) all the time. The PCS yields a total score and three subscale scores assessing rumination, magnification and helplessness. The PCS total score is computed by summing responses to all 13 items.
  PCS total scores range from 0 - 52 with higher scores indicating higher catastrophizing
Change in Depression | before surgery and 12 weeks post surgery
  Patient Health Questionnaire (PHQ-): 9-item depression questionnaire. Nine items, each of which is scored 0 to 3, providing a 0 to 27 severity score. Scores of 0-4 suggest no depression; Scores of 5-9 suggest mild depression; scores of 10-14 suggest moderate depression; scores of 15-19 suggest moderate-severe depression; scores of 20-27 suggest severe depression
Change in PROMIS (Patient-Reported Outcomes Measurement Information System) Global Health Scale | before surgery and 12 weeks post surgery
  The PROMIS Global-10 short form consists of 10 items that assess general domains of health and functioning including overall physical health, mental health, social health, pain, fatigue, and overall perceived quality of life. Participant's measures are reported as a transformed scale (or T-score). A higher PROMIS T-score represents more of the concept being measured
Change in Opioid Use | immediately after the intervention, 12 weeks post surgery
  Patient self reported: 1)opioid type; 2) surgical opioids yes/no; 3) total mg in past 24 hours; more than prescribed yes/no
Change in PROMIS Pain Interference | before surgery and 12 weeks post surgery
  This scale measures the construct of pain interference. Pain interference refers to the degree to which pain limits or interferes with an individual's physical, mental, and social activities. PROMIS Pain Interference scores are reported as a transformed scale (or T-score). A higher PROMIS T-score represents more of the concept being measured

CONTACTS AND LOCATIONS:
Overall Officials: Sara Davin, PsyD, MPH, Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic Foundation, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No